CLINICAL TRIAL: NCT05526924
Title: A Phase I Trial of Re-Irradiation With Concurrent Chemotherapy in Combination With Tislelizumab and Pamiparib in Patients With Previously Treated Head and Neck Squamous Cell Carcinoma
Brief Title: Dosing Study of Radiation Combined With Tislelizumab and Pamiparib in Patients With Previously Treated Head and Neck Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB22-0578
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma; Head and Neck Carcinoma; Head and Neck Cancer Stage IV; Head and Neck Cancers - Throat
Keywords: head and neck cancer; head and neck carcinoma; Head and Neck Squamous Cell Carcinoma; throat cancer; HNSCC treatment
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Chemoradiotherapy; pamiparib; Hydroxyurea; Fluorouracil; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose-Finding Group 1: Dose Level 1 (Part 1 of Study) (Experimental): The purpose of part 1 is to determine the best tolerated dose of study drugs with the least side effects. Dose escalation means that some participants will receive a different (higher) dose than other participants depending on when they join the study. This is to determine side effects at different doses and find a dose that will be safe to give to all participants. Participants in this group will receive:
  1. One dose of tislelizumab (200 mg) 15 days before chemoradiotherapy (CRT) given intravenously (by IV), which means through a vein.
  2. Chemoradiotherapy over a period of 5 weeks. During each cycle of CRT, participants will receive:
     * Pamiparib (20 mg daily on days 0-5 of each cycle) along with 5FU and hydroxyurea for 5 days.
     * Radiation will also be given two times a day for 5 days
  3. After CRT, participants will rest for roughly 8 days without study drugs or radiation then they will receive tislelizumab (200 mg) for 12 months by IV over 30 minutes every 6 weeks.
  Interventions: Radiation: Chemoradiation; Drug: Pamiparib; Drug: Hydroxyurea; Drug: Fluorouracil (5FU); Drug: Tislelizumab
- Dose-Finding Group 2: Dose Level 2 (Part 1 of Study) (Experimental): The purpose of part 1 is to determine the best tolerated dose of study drugs with the least side effects. Dose escalation means that some participants will receive a different (higher) dose than other participants depending on when they join the study. This is to determine side effects at different doses and find a dose that will be safe to give to all participants. Participants in this group will receive:
  1. One dose of tislelizumab (200 mg) 15 days before chemoradiotherapy (CRT) given intravenously (by IV), which means through a vein.
  2. Chemoradiotherapy over a period of 5 weeks. During each cycle of CRT, participants will receive:
     * Pamiparib (20 mg twice daily on days 0-5 of each 14 -day cycle) along with 5FU and hydroxyurea for 5 days.
     * Radiation will also be given two times a day for 5 days
  3. After CRT, participants will rest for roughly 8 days without study drugs or radiation then they will receive tislelizumab (200 mg) for 12 months by IV over 30 minutes every 6 weeks.
  Interventions: Radiation: Chemoradiation; Drug: Pamiparib; Drug: Hydroxyurea; Drug: Fluorouracil (5FU); Drug: Tislelizumab
- Dose-Finding Group 3: Dose Level 3 (Part 1 of Study) (Experimental): The purpose of part 1 is to determine the best tolerated dose of study drugs with the least side effects. Dose escalation means that some participants will receive a different (higher) dose than other participants depending on when they join the study. This is to determine side effects at different doses and find a dose that will be safe to give to all participants. Participants in this group will receive:
  1. One dose of tislelizumab (200 mg) 15 days before chemoradiotherapy (CRT) given intravenously (by IV), which means through a vein.
  2. Chemoradiotherapy over a period of 5 weeks. During each cycle of CRT, participants will receive:
     * Pamiparib (40 mg twice daily on days 0-5 of each 14 -day cycle) along with 5FU and hydroxyurea for 5 days.
     * Radiation will also be given two times a day for 5 days
  3. After CRT, participants will rest for roughly 8 days without study drugs or radiation then they will receive tislelizumab (200 mg) for 12 months by IV over 30 minutes every 6 weeks.
  Interventions: Radiation: Chemoradiation; Drug: Pamiparib; Drug: Hydroxyurea; Drug: Fluorouracil (5FU); Drug: Tislelizumab
- Dose Expansion Group ( Part II of Study) (Experimental): Part 2 (dose expansion phase): The purpose of this part is to continue to evaluate the dose of study drugs that is the best tolerated and has the least side effects. This part will start once the dose is selected from part 1. Enrollment in this part of the study is dependent on when participants join the study. Approximately 18 subjects will be enrolled in Part 2.
  Interventions: Radiation: Chemoradiation; Drug: Pamiparib; Drug: Hydroxyurea; Drug: Fluorouracil (5FU); Drug: Tislelizumab

INTERVENTIONS:
Radiation: Chemoradiation — A combination of chemotherapy and radiation given at the same time to treat cancer.
Drug: Pamiparib — An anti-cancer drug that targets specific cells to help fight cancer given by IV (through a needle inserted into a vein).
  Other Names: BGB-290
Drug: Hydroxyurea — A chemotherapy drug given in pill form; used to treat leukemia and head and neck cancer.
  Other Names: Hydrea; Droxia
Drug: Fluorouracil (5FU) — A chemotherapy drug used to treat different types of cancer.
  Other Names: Tolak; Fluoroplex; Efudex
Drug: Tislelizumab — An anti-cancer drug.
  Other Names: BGB-A317

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and maximum tolerated dose of tislelizumab in combination with pamiparib plus chemoradiotherapy (chemotherapy and radiation) in individuals with recurrent head and neck cancer, which means that the person's cancer has come back after treatment.

Participation in the study should last for about 15 months while participants receive tislelizumab and chemoradiotherapy with pamiparib. Afterwards, they will return to the clinic for follow up every 4 months for 2 years, every 6 month for the next 2 years, and then once a year for the rest of their life.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability and maximum tolerated dose of tislelizumab in combination with pamiparib plus chemoradiotherapy (chemotherapy and radiation) in individuals with recurrent head and neck cancer, which means that the person's cancer has come back after treatment.

During the study, participants will first receive one dose of tislelziumab. Tislelzumab is an experimental drug, meaning, it is not approved by the U.S. Food and Drug Administration (FDA) to treat cancer. Next, participants will receive pamiparib in combination with CRT (chemotherapy and radiation). Pamiparib is also an experimental drug and not approved by the FDA.

Chemoradiotherapy will consist of chemotherapy drugs, 5-FU and hydroxyurea, plus radiation therapy. 5-FU is approved by the FDA to treat many types of cancer such as colon cancer but has not been approved for the treatment of head and neck cancer. Its use is experimental in this study. Hydroxyurea is approved by the FDA to treat many types of cancer, including in combination with radiation therapy for the local control of squamous carcinoma of the head and neck. The combination of tislelizumab, hydroxyurea with 5-FU, radiation, and pamiparib, is considered experimental in this study.

Participation in the study should last for about 15 months while participants receive tislelizumab and chemoradiotherapy with pamiparib. Afterwards, they will return to the clinic for follow up every 4 months for 2 years, every 6 month for the next 2 years, and then once a year for the rest of their life.

ELIGIBILITY:
Inclusion Criteria:

* Clinically documented recurrent head and neck cancer requiring regional therapy.
* Human papillomavirus (HPV) testing for oropharynx primary tumors by p16 immunohistochemistry (IHC) positivity
* Availability of more than (or equal to) 10 unstained 5 micron slides (to be provided to Human Tissue Resource Center at the University of Chicago). Subjects who cannot fulfill this requirement will need to undergo a new biopsy prior to enrollment on study.
* Recurrent or second primary, previously irradiated head and neck squamous cell carcinoma without clinically measurably distant metastatic disease, or low volume oligometastatic disease amenable to Stereotactic Body Radiation Therapy (SBRT) or other curative-intent therapy (e.g. surgery, radiation frequency ablation therapy)
* Prior radiation therapy completed in 4 months (or longer) , and/or chemotherapy, immunotherapy, or targeted therapy completed 1 month (or earlier) before study entry, and patient should have recovered from any adverse effects.
* Prior programmed death-1 (PD-1)/ programmed death ligand-1 (PD-L1) inhibition is permitted.
* Prior chemotherapy is permitted.
* Patients who undergo surgical salvage therapy with positive margin or extranodal extension or other high-risk patients determined during multidisciplinary tumor board who are eligible for adjuvant re-irradiation therapy are eligible.
* 18 years of age and older.
* Eastern Cooperative Oncology Group performance status of one or less.
* Life expectancy of greater than 12 weeks.
* Negative serum or urine pregnancy test at screening for patients of childbearing potential.
* Patients must have normal organ and marrow functions as defined by lab values that will be confirmed by the study doctor.
* Age, Sex, and Reproductive Status:

  1. Women of childbearing potential (WOCBP=premenopausal woman capable of becoming pregnant) must have a negative serum or urine pregnancy test within 24 hours prior to the start of study drug.
  2. Women must not be breastfeeding.
  3. WOCBP must agree to follow instructions for highly effective method(s) of contraception for the duration of treatment and for 180 days (6 months) after the last dose of study drug(s).
  4. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 180 days (6 months) after the last dose of study drug(s).
  5. Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. Females must still undergo pregnancy testing as described in this section.

Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of <1% when used consistently and correctly.

* At a minimum subjects must agree to the use of one method of highly effective contraception as listed in Appendix D. In addition, male subjects are expected to use a condom as noted in Appendix D. The effects of tislelizumab and pamiparib on the developing human fetus are unknown. For this reason and because monoclonal antibodies and PARP inhibitor agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of pamiparib and tislelizumab administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* • Previously untreated patients with locoregional-only disease are not eligible.

  * Patients who have had chemotherapy within 4 weeks prior to entering the study, or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
  * Patients may not be receiving any other investigational agents.
  * History of allergic reactions attributed to compounds of similar chemical composition or excipients used in the study.
  * Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before the first dose of study drug(s).

    * Note: Patients who are currently or have recently been on any of the following corticosteroid regimens are not excluded:
* Adrenal replacement corticosteroid (dose ≤ 10 mg daily of prednisone or equivalent)
* Topical, ocular, intra-articular, intranasal, or inhalational corticosteroid with minimal systemic absorption
* Short course (≤ 7 days) of corticosteroid prescribed prophylactically (e.g., for contrast dye allergy) or for the treatment of a nonautoimmune condition (e.g., delayed-type hypersensitivity reaction caused by contact allergen)

  * Has hypersensitivity to tislelizumab, pamiparib, or any other drug used in this protocol.
  * Has a known history of active tuberculosis (Bacillus Tuberculosis infection)
  * Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer or any tumors that are not likely to influence live expectancy in the subsequent 3 years without active treatment (e.g. low grade prostate cancer in absence of therapy), or prior history of acute myeloid leukemia (AML)/myelodysplastic syndrome (MDS).
  * Has active autoimmune disease that has required systemic treatment in the past year (i.e. with use of steroids or immunosuppressive drugs). Replacement therapy e.g. levothyroxine, insulin, or physiologic corticosteroid doses for adrenal or pituitary insufficiency, etc. are not considered a form of systemic treatment.
  * Has known history of, or any evidence of active interstitial lung disease, noninfectious pneumonitis, or uncontrolled lung diseases including pulmonary fibrosis, or acute lung diseases.
  * Has a history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
  * Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected). However, if eradicated subject is eligible.
  * Has received a live vaccine within 28 days of planned start of study therapy.

    o Note: Vaccines for COVID-19 are allowed except for any live vaccine that may be developed. Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed within 28 days prior to initiation of treatment. Vaccines should not be given during the chemo-radiation phase until marrow function has normalized as vaccines may not be efficacious during periods of marrow suppression.
  * Uncontrolled intercurrent illness including but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
  * Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
  * Patients receiving any medications or substances that are known to be strong CYP3A inducers (eg. avasimibe, carbamazepine, mitotane, phenobarbital, phenytoin, rifabutin, rifampin/ rifampicin) are ineligible. Patients receiving herbal remedies/medicines such as St. John's Wort (Hypericum perforatum) are also ineligible. See Sections 5.5.2 and 5.5.3 for prohibited medications on study.

Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.

* Pregnant women are excluded from this study because pamiparib is a PARP inhibitor and tislelizumab is a humanized, immunoglobulin G4 (IgG4)-variant monoclonal antibody agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pamiparib and tislelizumab, breastfeeding should be discontinued if the mother is treated with pamiparib and tislelizumab.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with pamiparib and tislelizumab. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Disease/procedure significantly affecting gastrointestinal function, such as malabsorption syndrome, resection of the stomach or small bowel, bariatric surgery procedures, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction, or gastrointestinal perforation or fistulae. Note: Gastroesophageal reflux disease under treatment with proton pump inhibitors is allowed (assuming no drug interaction potential).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose/Recommended Phase 2 Dose of Pamiparib in Combination with 5 Fluorouracil-Hydroxea (FHX) and Tislelizumab | 15 months
  Determine the maximally tolerated dose (MTD)/ recommended phase 2 dose (RP2D) for pamiparib in combination with FHX and tislelizumab in subjects with recurrent head and neck squamous cell carcinoma (HNSCC) as assessed by the incidence of dose-limiting toxicities (side effects) reported among study participants. Dose-limiting toxicities will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.

SECONDARY OUTCOMES:
Progression Free Survival of Participants Receiving Pamiparib in Combination with 5 Fluorouracil-Hydroxea (FHX) and Tislelizumab | 15 months
  The progression free survival (PFS) of participants receiving pamiparib in combination with FHX and tislelizumab in subjects with recurrent head and neck squamous cell carcinoma, defined as the time from initiation of treatment with tislelizumab to the earliest of disease progression per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) or death from any cause.
Overall Free Survival of Participants Receiving Pamiparib in Combination with 5 Fluorouracil-Hydroxea (FHX) and Tislelizumab | 15 months
  Overall survival (OS) of participants receiving pamiparib in combination with FHX and tislelizumab in subjects with recurrent head and neck squamous cell carcinoma, defined as the time from initiation of treatment with tislelizumab to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ari Rosenberg, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes